CLINICAL TRIAL: NCT04862039
Title: Use of Virtual Reality in Active Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, PI MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 485/20
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) devices (Experimental): intervention group (VR).
  Interventions: Device: Virtual Reality (VR) devices
- control group (No Intervention): the standard of care (control group, no VR)

INTERVENTIONS:
Device: Virtual Reality (VR) devices — Virtual Reality (VR) devices. Subjects receiving the experimental treatment will be given a VR headset, headphones and wristband and the Philips wireless fetal-maternal monitoring system, after the necessary preparation of the abdominal skin.
  Arms: Virtual Reality (VR) devices

SUMMARY:
Labor is widely recognized as one of the most painful experience possible. The standard analgesic treatment currently consists of pharmacological methods. Adverse effects, complication risks, psychological effects, limit these techniques as well as high costs. These limits concurred to the application of these techniques mainly on demand and not routinely. have not, as of today, met a large scientific consensus, as shown by many recent Cochrane reviews. A promising perspective for non-pharmacological analgesia seems to be offered by Virtual Reality (VR) devices, which have been applied to many different medical areas.

DETAILED DESCRIPTION:
Labor is widely recognized as one of the most painful experience possible. The standard analgesic treatment currently consists of pharmacological methods. Adverse effects, complication risks, psychological effects, limit these techniques as well as high costs. These limits concurred to the application of these techniques mainly on demand and not routinely.

For all these reasons, it is not surprising the interest in offering women valid non-invasive and cheaper options to relieve them from pain. As of today many alternative techniques have been proposed, many of which have not, as of today, met a large scientific consensus, as shown by many recent Cochrane reviews. A promising perspective for non-pharmacological analgesia seems to be offered by Virtual Reality (VR) devices, which have been applied to many different medical areas. Recently Frey et al. have experimented in a pilot study the application of this technique to women during labor, obtaining interesting results. The authors of this study point, in the discussion of the scientific paper, to the necessity of developing virtual reality experiences more specific to labor and suggest different implementations, such as specific instructions for women (changes of position, breathing techniques) greater comfort (it is worth noticing the use on our side of exclusively wireless devices) and the implementation of the device with biofeedback.

In addition to learning from these suggestions, we tried to imagine VR in a different way: firstly as complementary, not alternative to the role of the midwife personnel, who will play a central role in our experimental treatment enriching the virtual reality scenario with their instructions, presence and motivational feedback; secondly we tried to imagine VR as a guide through labor, more than a alienation and distraction tool.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestations;
* term pregnancy
* spontaneous labor
* diagnosis of active phase of labor;
* nulliparous between 37 and 42 gestation weeks with cephalic presentation ;

Exclusion Criteria:

* multiple gestations;
* preterm labor;
* preterm premature rupture of membranes
* induction to delivery labor;
* hipertensive disorders;
* fetal abnormalities;
* diabetes mellitus;
* intrauterine growth retardation;
* post-term pregnancy;
* multiple vaginal delivery;
* women with an altered state of consciousness, severely ill, mentally disabled;
* women with sight and/or hearing impairment;
* women at risk of epileptic seizures;
* women with predisposition to motion sickness;
* women under the age of 18 years or over the age of 45 years;
* Women who refuse to sign informed informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Subjective pain during the active phase | "during the active phase of labor up to 10 cm"
  women pain using visual analogue scale (VAS)

SECONDARY OUTCOMES:
nausea | during the active phase of labor (i.e. after 4-6 cm of dilatation)
  nausea referred by the patient and episodes of vomiting
anxiety | during the active phase of labor (i.e. after 4-6 cm of dilatation)
  women axneity using visual analogue scale (VAS)
Incidence of episiotomy | at the time of delivery
  Incidence of episiotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Naples, Italy

IPD SHARING:
Plan to Share IPD: No
none planned